CLINICAL TRIAL: NCT04779359
Title: The Predictive Role of Lymphocyte Subsets and Laboratory Measurements in COVID-19 Disease- A Retrospective Study
Brief Title: Role of Lymphocyte Subsets and Laboratory Measurements in COVID-19 Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Public Health Clinical Center (Other Government)
Responsible Party: Principal Investigator, Hongzhou Lu, • Co-Director of Shanghai Public Health Clinical Center affiliated to Fudan University, Shanghai Public Health Clinical Center
Other Study IDs: COVID-19 Disease
Record Dates: First submitted 2021-03-01; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: COVID-19 Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate the predictive role of lymphocyte subsets and other laboratory measurements in adult patients with COVID-19.This was a single center, retrospective study that involved adult patients with confirmed diagnosis of COVID-19. Electronic medical records were reviewed. Data including age, sex, symptom from onset to hospital admission and laboratory findings at admission of hospitalized patients with confirmed COVID-19 were extracted and analyzed retrospectively.This study indicates that the levels of lymphocyte subsets (CD4+, and CD8+) are associated with disease progression and severity, along with prognosis in patients with COVID-19.

DETAILED DESCRIPTION:
This was a single center, retrospective study that involved adult patients with confirmed diagnosis of COVID-19. Electronic medical records were reviewed. Data including age, sex, symptom from onset to hospital admission and laboratory findings at admission of hospitalized patients with confirmed COVID-19 were extracted and analyzed retrospectively. Identifying the possible immune factors and laboratory parameters is requisite for the early identification of patients with severe COVID-19 and timely intervention for control of the disease. There is an unmet need to establish robust clinical cutoffs of lymphocyte subsets for predicting risk associated with ICU admission, mechanical ventilation, and mortality in COVID-19 patients. This retrospective study was thus carried out to improve knowledge and clinical utility of lymphocyte subset measurements, together with other laboratory measurements and clinical information, for understanding prognosis in COVID-19 patients. These findings suggest that alterations in lymphocyte subsets and laboratory measurements play a significant role in the progression of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of COVID-19 disease.

Exclusion Criteria:

* The patients were excluded patients <18 years age and without confirmed diagnosis of disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients were included for this study after excluding patients <18 years age and without confirmed diagnosis of disease.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Correlation of CD4+ and CD8+ T cell absolute counts to disease outcomes | 2021.02-2021.08
  The study endpoints were to demonstrate whether CD4+ and CD8+ T cell absolute counts are prognostic marker in determining disease outcomes (including ICU admission and/or mechanical ventilation and/or mortality); to explore whether lymphocyte subset measurements recover at hospital discharge or in convalescence; lymphocyte subset measurements between severe and non-severe groups, at admission. In addition, association between CD4+ and CD8+ T cell absolute counts with cytokine levels and other laboratory parameters (neutrophil counts, total lymphocyte counts, platelet counts, C-reactive protein levels) were also assessed.